CLINICAL TRIAL: NCT01125605
Title: PASCONAL NERVENTROPFEN in the Treatment of Adults and Children Suffering From Nervous Diseases (e.g. Sleep Disorders Due to Nervousness)
Brief Title: PASCONAL NERVENTROPFEN in the Treatment of Nervous Diseases
Acronym: 174
Status: Completed | Type: Observational
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 174A10PNAL
Record Dates: First submitted 2010-05-10; First posted 2010-05-18 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Nervousness; Sleep Disorders
Keywords: PASCONAL; nervousness; nervosity; sleep disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Adults > 12 years: adult patients and patients older than 12 years
- Children 6-12 years: children between 6 and 12 years
- Children 1-6 years: children between 1 and 6 years

SUMMARY:
The purpose of this observational study is to give an overview of the use of PASCONAL NERVENTROPFEN in a 2-4 week treatment of nervous diseases, especially sleep disorders due to nervousness.

DETAILED DESCRIPTION:
The purpose of this observational study is to give an overview of the use of PASCONAL NERVENTROPFEN in a 2-4 week treatment of nervous diseases, especially sleep disorders due to nervousness.

Efficacy and tolerability of the drug will be assessed. Special regard will be taken to the administration management, dose regimen, and to the effectiveness and safety in special patient groups (children 1-12 years of age), in relation to treatment conformity to the Summary of Product Characteristics (SmPC).

ELIGIBILITY:
Due to the design as an Observational Study no inclusion or exclusion criteria for therapy are named. The included patient group is described under "Cohort / Group".

Observational Criteria (=inclusion criteria for documentation):

* Males and females
* Children 1-12 years old
* Adults >12 years old
* suffering from nervous diseases, e.g. sleep disorders due to nervousness.

Exclusion criteria for documentation:

* children younger than 1 year
* no nervous diseases, e.g. sleep disorders due to nervousness.
* no treatment with PASCONAL NERVENTROPFEN

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Observational groups
  Patients (adults and children 1-12 years of age) suffering from nervous diseases, e.g. sleep-disturbances due to nervousness.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bianka Krick, Study Director — Pascoe Pharmazeutische Praeparate GmbH
Locations (1):
- Multiple German Practices, All Over Germany, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Physicians who were registered in the past with the treatment focus on central nervous system / psyche. The recruitment of the participating physicians was done by the field service of PASCOE.
Pre-assignment Details: It was an non-inteventional observational study with 3 visits.
Groups:
- Observational Group: Pasconal Nerventropfen PASCONAL® NERVENTROPFEN is a homoeopathic combination product (oral drops) consisting out of 4 ingredients: Avena sativa, Valeriana, Ignatia and Tarantula.
Period: Overall Study
Arm/Group | Observational Group
Started | 325 (started = had baseline values)
Safety | 326 (1 patient was only analysed for safety)
Completed | 325
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Observational Group: Pasconal Nerventropfen
Arm/Group | Observational Group
Number analyzed (Participants) | 325
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 72
  Between 18 and 65 years | 212
  >=65 years | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229
  Male | 96
Concomitant medication [Number; unit: participants]
  with concomitant medication | 176
  without concomitant medication | 149
Duration of disease years [Mean (Standard Deviation); unit: years] | 2.0 (3.8)
State of inclusion diagnosis [Number; unit: participants] — The duration of complaints was divided into two groups to the extent this was possible:
  * Acute disease (duration of symptoms ≤2 months)
  * Subchronic and/or chronic disease (duration of symptoms >2 months)
  participants
    acute (<= 2 months) | 43
    subchronic/chronic (> 2 months) | 163
    missing data | 119
Previous treatment of inclusion diagnosis [Number; unit: participants] — Within the range of the observational study, it was ascertained whether the inclusion diagnosis had been treated previously.
  participants
    with previous treatment of inclusion diagnosis | 245
    without previous treatment of inclusion diagnosis | 80

OUTCOME MEASURES:

1. Primary Outcome: Sumscore of 12 Individual Symptoms for Visit 1 (Baseline), Visit 2, and Visit 3
Description: The severity of 12 symptoms (nervousness/restlessness, irritability/eccentricity, sleep disorders, fitful sleep, hyperactivity, nocturnal activity, lack of concentration/forgetfulness, tiredness, discontent, listlessness, gastrointestinal problems, and headache/pressure) was graded on a four-point scale from 0 (no complaints) to 3 (strong complaints) and for the sum score of all 12 individual symptom scores (0 (no complaints) - 36 (all strong complaints).
Time Frame: begin (visit 1), appr. after 2 weeks (visit 2), and appr. after 4 weeks (visit 3)
Population: descriptive; for all partcipations with values at the visits
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Visit 1: Observational group (Pasconal Nerventropfen) at visit 1
- Visit 2: Observational group (Pasconal Nerventropfen) at visit 2
- Visit 3: Observational group (Pasconal Nerventropfen) at visit 3
- Last Observation: Observational group (Pasconal Nerventropfen) at last observation
Arm/Group | Visit 1 | Visit 2 | Visit 3 | Last Observation
Number analyzed (Participants) | 325 | 325 | 309 | 325
units on a scale | 15.8 (6.1) | 9.2 (5.6) | 5.1 (4.5) | 6.2 (5.2)

2. Secondary Outcome: Changes of the Sum Score Between Baseline and Last Observation by Concomitant Medication and Treatment Duration
Description: The severity of 12 symptoms (nervousness/restlessness, irritability/eccentricity, sleep disorders, fitful sleep, hyperactivity, nocturnal activity, lack of concentration/forgetfulness, tiredness, discontent, listlessness, gastrointestinal problems, and headache/pressure) was graded on a four-point scale from 0 (no complaints) to 3 (strong complaints) and for the sum score of all 12 individual symptom scores (0 (no complaints) - 36 (all strong complaints).
  Decrease of the sumscore between baseline and last observation by concomitant medication (with and withour medication) and treatment duration (< 4 weeks and >= 4 weeks)
Time Frame: begin (visit 1) and last obvservation (could be appr. after 2 weeks (visit 2) or 4 weeks (visit 3))
Population: exploratively, all participations with values
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Visit 1 | Last Observation
Number analyzed (Participants) | 325 | 325
units on a scale
  with concomitant medication | 15.9 (5.5) | 7.7 (5.6)
  without concomitant medication | 15.7 (6.2) | 5.8 (5.0)
  < 4 weeks treatment duration | 14.3 (5.3) | 7.4 (6.0)
  >= 4 weeks treatment duration | 16.1 (6.2) | 5.9 (4.9)
Statistical Analysis 1: Comparison: Visit 1 vs Last Observation; decrease of the sum score between baseline (visit 1) and last observation was exploratively analysed; Test type: Superiority or Other; p = 0.0033, ANCOVA; ANCOVA with GLM (Generalized Linear Model) of SAS® (with type III sums of squares); including the baseline value of the sum score as a covariate
Statistical Analysis 2: Comparison: Visit 1 vs Last Observation; decrease of the sum score between baseline (visit1) and last observation by duration of treatment; Test type: Superiority or Other; p = 0.0002, ANCOVA; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Direction of Change of Symptom Nervousness/Restlessnes Between Baseline and Last Observation by Concomitant Medication
Description: The symptom nervousness/restlessnesswas analysed with respect to the direction of change between baseline (Visit 1) and the last documented visit (Visit 2 or Visit 3) by means of the categories "improved", "unchanged" and "worsened". For each symptom patients were included in the analysis only if the symptom had been present at Visit 1 (i.e. the baseline score value was > 0).
Time Frame: begin (visit 1) and last observation (could be appr. after 2 weeks (visit 2) or appr. after 4 weeks (visit 3))
Population: exploratively, all participations with values
Measure: Number; unit: participants
Groups:
- With Concomitant Medication: Observational group (Pasconal Nerventropfen) with concomitant medication
- Without Concomitant Medication: Observational group (Pasconal Nerventropfen) without concomitant medication
Arm/Group | With Concomitant Medication | Without Concomitant Medication
Number analyzed (Participants) | 68 | 240
participants
  improved | 46 | 206
  unchanged | 19 | 32
  worsened | 3 | 2
Statistical Analysis 1: Comparison: With Concomitant Medication vs Without Concomitant Medication; Test type: Superiority or Other; p = 0.0014, Fisher Exact

4. Secondary Outcome: Direction of Change of Symptom Nervousness/Restlessnes Between Baseline and Last Observation by Duration of Treatment
Description: The symptom nervousness/restlessness was analysed with respect to the direction of change between baseline (Visit 1) and the last documented visit (Visit 2 or Visit 3) by means of the categories "improved", "unchanged" and "worsened". For each symptom patients were included in the analysis only if the symptom had been present at Visit 1 (i.e. the baseline score value was > 0).
Time Frame: begin (visit 1) and last observation (could be appr. after 2 weeks (visit 2) or appr. after 4 weeks (visit 3))
Population: exploratively, all participations with values
Measure: Number; unit: participants
Groups:
- < 4 Weeks: Observational group (Pasconal Nerventropfen) with a treatment duration < 4 weeks
- > = 4 Weeks: Observational group (Pasconal Nerventropfen) with a treatment duration >= 4 weeks
Arm/Group | < 4 Weeks | > = 4 Weeks
Number analyzed (Participants) | 65 | 243
participants
  improved | 46 | 206
  unchanged | 16 | 35
  worsened | 3 | 2
Statistical Analysis 1: Comparison: < 4 Weeks vs > = 4 Weeks; Test type: Superiority or Other; p = 0.0125, Fisher Exact

5. Secondary Outcome: Direction of Change of Symptom Irritability/Eccentricity Between Baseline and Last Observation by Concomitant Medication
Description: The symptom irritability/eccentricity was analysed with respect to the direction of change between baseline (Visit 1) and the last documented visit (Visit 2 or Visit 3) by means of the categories "improved", "unchanged" and "worsened". For each symptom patients were included in the analysis only if the symptom had been present at Visit 1 (i.e. the baseline score value was > 0).
Time Frame: begin (visit 1) and last observation (could be appr. after 2 weeks (visit 2) or appr. after 4 weeks (visit 3))
Population: exploratively, all participations with values
Measure: Number; unit: participants
Arm/Group | With Concomitant Medication | Without Concomitant Medication
Number analyzed (Participants) | 66 | 227
participants
  improved | 43 | 195
  unchanged | 21 | 30
  worsened | 2 | 2
Statistical Analysis 1: Comparison: With Concomitant Medication vs Without Concomitant Medication; Test type: Superiority or Other; p = 0.0006, Fisher Exact

6. Secondary Outcome: Direction of Change of Symptom Irritability/Eccentricity Between Baseline and Last Observation by Duration of Treatment
Description: as for outcome 5
Time Frame: begin (visit 1) and last observation (appr. after 2 weeks (visit 2) or appr. after 4 weeks (visit 3))
Population: exploratively, all participations with values
Measure: Number; unit: participants
Arm/Group | < 4 Weeks | > = 4 Weeks
Number analyzed (Participants) | 61 | 232
participants
  improved | 40 | 198
  unchanged | 19 | 32
  worsened | 2 | 2
Statistical Analysis 1: Comparison: < 4 Weeks vs > = 4 Weeks; Test type: Superiority or Other; p = 0.0016, Fisher Exact

7. Secondary Outcome: Efficacy Rating for PASCONAL® NERVENTROPFEN (Last Value) Compared to Previous Therapy by Concomitant Medication (Yes/no)
Description: Efficacy of the therapy with PASCONAL® NERVENTROPFEN was rated by the physician on a 4-point rating scale at Visit 2 and Visit 3. The same scale was applied at Visit 1 for evaluation of the efficacy of the previous medication.
  The last evaluation for PASCONAL® NERVENTROPFEN (Visit 2 or Visit 3, according to the LOCF principle) was compared with the rating for the previous therapy by means of the categories "PASCONAL® better", "No difference" and "PASCONAL® worse".
Time Frame: appr. after 2 weeks (visit 2) and appr. after 4 weeks (visit 3)
Population: exploratively, all participations with values
Measure: Number; unit: participants
Arm/Group | With Concomitant Medication | Without Concomitant Medication
Number analyzed (Participants) | 68 | 174
participants
  PASCONAL better | 40 | 128
  No difference | 18 | 34
  PACONAL worse | 10 | 12
Statistical Analysis 1: Comparison: With Concomitant Medication vs Without Concomitant Medication; Test type: Superiority or Other; p = 0.0504, Fisher Exact

8. Primary Outcome: Nervousness/Restlessness for Visit 1 (Baseline), Visit 2, Visit 3 and Last Obsevation
Description: The severity of nervousness/restlessness was graded on a four-point scale from 0 (no complaints) to 3 (strong complaints).
Time Frame: begin (visit 1), appr. after 2 weeks (visit 2), and appr. after 4 weeks (visit 3)
Population: descriptive; for all partcipations with values at the visits
Measure: Number; unit: participants
Groups:
- Visit 3: Observational group (Pasconal Nerventropfen) at visit 1
Arm/Group | Visit 1 | Visit 2 | Visit 3 | Last Observation
Number analyzed (Participants) | 308 | 306 | 293 | 308
participants
  0=not present | 0 | 23 | 78 | 79
  1=mild | 63 | 171 | 180 | 789
  2=moderate | 166 | 98 | 26 | 29
  3=Strong | 79 | 14 | 9 | 11

9. Secondary Outcome: Efficacy Rating for PASCONAL® NERVENTROPFEN (Last Value) Compared to Previous Therapy by Treatment Duration
Description: as for outcome 7
Time Frame: appr. after 2 weeks (visit 2) and appr. after 4 weeks (visit 3)
Population: exploratively, all participations with values
Measure: Number; unit: participants
Groups:
- < 4 Weeks: Observational group (Pasconal Nerventropfen) with concomitant medication
- >= 4 Weeks: Observational group (Pasconal Nerventropfen) without concomitant medication
Arm/Group | < 4 Weeks | >= 4 Weeks
Number analyzed (Participants) | 52 | 190
participants
  PASCONAL better | 25 | 143
  No difference | 16 | 36
  PACONAL worse | 11 | 11
Statistical Analysis 1: Comparison: < 4 Weeks vs >= 4 Weeks; Test type: Superiority or Other; p = 0.0002, Fisher Exact

10. Primary Outcome: Irritability/Eccentricity for Visit 1 (Baseline), Visit 2, Visit 3 and Last Observation
Description: The severity of irritability/eccentricity was graded on a four-point scale from 0 (no complaints) to 3 (strong complaints).
Time Frame: begin (visit 1), appr. after 2 weeks (visit 2), and appr. after 4 weeks (visit 3)
Population: descriptive; for all partcipations with values at the visits
Measure: Number; unit: participants
Arm/Group | Visit 1 | Visit 2 | Visit 3 | Last Observation
Number analyzed (Participants) | 293 | 291 | 278 | 293
participants
  0=not present | 0 | 41 | 111 | 115
  1=mild | 86 | 163 | 136 | 142
  2=moderate | 140 | 72 | 25 | 27
  3=Strong | 67 | 15 | 6 | 9

11. Primary Outcome: Tolerability After Visit 2 and Visit 3
Description: Assessment of tolerability at visit 2 and visit 3 well tolerated = no side effcts poor tolerated = side effects
Time Frame: appr. after 2 weeks (visit 2), and appr. after 4 weeks (visit 3)
Population: descriptive; for safety 326 patients were analysed; 1 patient had no efficacy values and were not analysed for efficacy; so a discrepancy between 325 patients (for efficacy) and 326 (for safety) occured
Measure: Number; unit: participants
Arm/Group | Visit 2 | Visit 3
Number analyzed (Participants) | 326 | 326
participants
  well tolerated | 313 | 303
  poor tolerated | 13 | 23

ADVERSE EVENTS:
Time Frame: after appr. 2 weeks and after appr. 4 weeks
Arm/Group | Observational Group
Serious Adverse Events (participants affected / at risk) | 0/326
Other Adverse Events (participants affected / at risk) | 14/326
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Group (N=326)
gastrointestinal (Gastrointestinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2)
tiredness (General disorders) | 3 (3)
headache (Nervous system disorders) | 2 (2)
tachycardia (Cardiac disorders) | 1 (1)
heartburn (Gastrointestinal disorders) | 1 (1)
aggressivity (Psychiatric disorders) | 1 (1)
stomach ache (Gastrointestinal disorders) | 1 (1)
tongue and mucosa under tongue (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes